CLINICAL TRIAL: NCT01542567
Title: Efficacy of Diclofenac Suppositories in Prevention of Immediate Side Effects of BCG Bladder Irrigations. A Double Blind Placebo Controlled Randomized Study
Brief Title: Efficacy of Diclofenac BCG Irrigations
Acronym: DIC-2011
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Avi Stein, M.D., Prof Avi Stein, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CMC-11-0015-CTIL
Record Dates: First submitted 2012-02-14; First posted 2012-03-02 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Bladder Cancer
Keywords: Diclofenac; BCG; BLADDER IRRIGATIONS
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- diclofenac (Active Comparator): suppositories to prevent BCG side effects
  Interventions: Drug: Abitren
- placebo suppositories (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abitren — SUPPOSITORIES 50 Mg 2 SUPPOSITORIES A WEEK
  Arms: diclofenac
Drug: Placebo — Placebo suppositories
  Arms: placebo suppositories

SUMMARY:
This study is designed to test the effectiveness of diclofenac suppositories in the prophylaxis of side effects caused by BCG bladder irrigations in bladder cancer patients.

DETAILED DESCRIPTION:
This study is designed as a double blind placebo controlled randomized study to evaluate the effectiveness of diclofenac suppositories in the prevention of side effects of BCG bladder irrigation in bladder cancer patients. After signing an informed consent, the patients will be randomized to either receive an unmarked suppository of Diclofenac or a placebo suppository. The effectiveness of the drug will be tested weekly by quality of life questionnaires and bladder symptom questionnaire. Another questionnaire is designed to monitor the time in minutes that the BCG is retained in the bladder before the patients urinates.

ELIGIBILITY:
Inclusion Criteria:

1. Bladder urothelial carcinoma patients scheduled fo a set of 6 BCG bladder irrigations at the Carmel Medical Centre
2. Male and female
3. Age 20-80.
4. Patients capable of understanding reading and signing the informed consent form in Hebrew.

Exclusion Criteria:

1. Diclofenac hypersensitivity
2. Pregnancy, Lactation
3. Elevated creatinine at baseline (male > 1.2 mg/% female 1.0 mg/%)
4. Peptic gastric or duodenal ulcer
5. Acute or chronic inflammation of the rectum/ anus (diarrhea, rectal bleeding)
6. Gross hematuria (which is per se a contraindication for BCG irrigation)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Change in weekly COOP Questionnaire 1 | The questionnaires will be completed every week for the quality of life of the passing week. The complete time frame of all questionnaires will be 7 weeks
  The bladder irrigations are delivered as an ambulatory treatment once a week. The questionnaires will be completed every week for the quality of life of the passing week.
Change in weekly COOP Questionnaire 2 | The questionnaires will be completed every week for the quality of life of the passing week. The complete time frame of all questionnaires will be 7 weeks
  The bladder irrigations are delivered as an ambulatory treatment once a week. The questionnaires will be completed every week for the quality of life of the passing week.
Change in weekly COOP Questionnaire 3 | The questionnaires will be completed every week for the quality of life of the passing week. The complete time frame of all questionnaires will be 7 weeks
  The bladder irrigations are delivered as an ambulatory treatment once a week. The questionnaires will be completed every week for the quality of life of the passing week.
Change in weekly Bladder symptoms Questionnaire | The questionnaires will be completed every week for the bladder symptoms of the passing week. The complete time frame of all questionnaires will be 7 weeks
  Bladder symptoms Questionnaire correlated to BCG treatment. The bladder irrigations are delivered as an ambulatory treatment once a week. The questionnaires will be completed every week for the bladder symptoms of the passing week.
Change in weekly time schedule questionnaire | every week for 6 weeks
  A questionnaire designed to measure the time in minutes that the patient was able to retain the BCG in the bladder.This questionnaire will be completed every week for the same day of weekly irrigation.